CLINICAL TRIAL: NCT03016598
Title: 6-week Trial of Oxytocin for Co-occurring Cocaine and Opioid Use Disorders
Brief Title: Stimulant Oxytocin Study
Acronym: SOS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NURA-014-16S; 1IK2CX001495-01 (NIH)
Record Dates: First submitted 2017-01-04; First posted 2017-01-10 (Estimated); Results first posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Stimulant Use & Co-occuring Opioid Use Disorders
Keywords: oxytocin; substance-related disorders; Opioid Replacement Therapy; Psychophysiology; Stress Biomarkers
MeSH Terms: conditions — Substance-Related Disorders | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxytocin (Experimental): Patients in methadone maintenance treatment (MMT) programs are required to come in every day for their methadone. Additionally they are required to come in weekly for psycho- educational/therapy groups, biweekly random urine screenings, and monthly individual therapy sessions. The investigators will piggy-back off this existing structure and randomize Veterans with stimulant use disorders and receiving MMT for co-occurring opioid use disorder (OUD) to receive either oxytocin or placebo, to be administered twice daily for six weeks while in the MMT program.
  Interventions: Drug: Intranasal oxytocin
- Placebo (Placebo Comparator): Patients in MMT programs are required to come in every day for their methadone. Additionally they are required to come in weekly for psycho- educational/therapy groups, biweekly random urine screenings, and monthly individual therapy sessions. The investigators will piggy-back off this existing structure and randomize Veterans with stimulant use disorders and receiving MMT for co-occurring OUD to receive either oxytocin or placebo, to be administered twice daily for six weeks while in the MMT program.
  Interventions: Drug: Intranasal placebo

INTERVENTIONS:
Drug: Intranasal oxytocin — Each Veteran with a stimulant use disorder, receiving MMT for OUD will receive a oxytocin nasal spray 40 International Units (IU) to be self administered twice daily over 6 weeks while in the MMT program. The veteran will come in for a total of 7 weekly visits. At baseline and during the last visit the veteran will complete at Trier Social Stress Test (TSST), and psychophysiological and biomarkers of stress will be collected. At every weekly visit a urine sample and self-reported drug use will be collected and therapy attendance will be recorded.
  Other Names: Syntocinon
  Arms: Oxytocin
Drug: Intranasal placebo — Each Veteran with a stimulant use disorder, receiving MMT for OUD will receive a placebo nasal spray 40IU to be self administered twice daily over 6 weeks while in the MMT program. The veteran will come in for a total of 7 weekly visits. At baseline and during the last visit the veteran will complete at Trier Social Stress Test (TSST), and psychophysiological and biomarkers of stress will be collected. At every weekly visit a urine sample and self-reported drug use will be collected and therapy attendance will be recorded.
  Other Names: Saline placebo
  Arms: Placebo

SUMMARY:
This study will investigate the effects of intranasal administration of oxytocin, a social neuropeptide, on reducing stimulant use, enhancing therapeutic engagement, and susceptibility to stress-induced relapse in Veterans with stimulant use disorders and enrolled in opioid replacement therapy (ORT) program for co-occurring opioid use disorder (OUD).

DETAILED DESCRIPTION:
High rates of substance use disorders (SUDs) in Veterans compared to the general population are heavily influenced by psychosocial factors - such as difficulty reintegrating into civilian life due to avoidance of vital support systems - leading to disproportionately elevated unmet addiction treatment needs. Although the gold standard for treatment for most SUDs involves pharmacological interventions, there are currently no effective pharmacological interventions approved by the Federal Drug Administration for stimulant users, who have the most difficulty adhering to treatment programs and the most susceptibility to stress-induced relapse of any SUD. Administering oxytocin, a mammalian neuropeptide, intranasally to healthy controls facilitates the stress-buffering properties of social support. Oxytocin may also have an independent role in mitigating the symptoms of SUDs. For example, in animal models of addiction, oxytocin administration directly reduces tolerance, withdrawal effects, self-administration, and stress-induced reinstatement of drug seeking for a range of addictive substances. A more integrated understanding of oxytocin's distinct effects on the behavior and psychology of 1) addiction, 2) sociality, and 3) stress reactivity could be the key to defining oxytocin's role in SUD treatment. This study proposes to translate promising preclinical and early proof-of-concept clinical results related to the anti-addiction, pro-social, and stress-tempering properties of oxytocin administration in Veterans with moderate-severe stimulant use disorders enrolled in a opioid replacement therapy (ORT) program for co-occurring opioid use disorder (OUD) at the San Francisco VA Medical Center (SFVAMC). The investigators' primary outcome is Aim 1) reduction in stimulant use, as measured by stimulant positive urine drug screen. Secondarily, the investigators will focus on Aim 2) improving psychosocial treatment engagement (social support) and Aim 3) mitigating social stress-related relapse, targeting two important barriers to stimulant use disorder recovery likely to respond to oxytocin administration.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old
2. Enrolled as a patient who at the SFVAMC Opioid Treatment Program or the Oakland Behavioral Health Clinic Opioid Treatment Program
3. Stable dose of opioid replacement therapy for at least 2 consecutive weeks
4. Veteran
5. One documented urine toxicology screen positive for stimulants in the past 12 months.

Exclusion Criteria:

1. Severe neuropsychological disorder
2. Suicidal or homicidal ideation within the past 90 days or a suicide attempt in the past 6 months
3. Hemodialysis, unless participant can produce urine samples weekly
4. Sensitivity to methylparaben or propylparaben
5. Positive urine pregnancy test or women of childbearing age not practicing effective means of non-hormonal birth control
6. Chronic nasal obstruction, discharge, or bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Stauffer, MD, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (3):
- United States (3):
  - VA Northern California Health Care System, Mather, CA, Sacramento, California
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California
  - VA Portland Health Care System, Portland, OR, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stauffer CS, Woolley JD. Can we bottle psychosocial treatments for addiction? The role of oxytocin. J Clin Psychiatry. 2014 Sep;75(9):1028-9. doi: 10.4088/JCP.14ac09437. No abstract available. PMID 25295428
- See also: Social Neuroscience & Psychotherapy Lab — https://www.chrisstauffermd.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 84 individuals assessed for eligibility, of which 38 were excluded. 28 of the 38 excluded were ineligible - 6 were lost to follow up and 4 were uninterested. The remaining 46 participants completed baseline assessment, of which 4 were excluded - 2 being ineligible, 1 being lost to follow up and the final being uninterested. Left remaining were 42 enrolled participants.
Pre-assignment Details: 42 individuals were enrolled, 2 of which were excluded due to being lost to follow up before being assigned to an arm.
Groups:
- Oxytocin: Patients in MMT programs are required to come in every day for their methadone. Additionally they are required to come in weekly for psycho- educational/therapy groups, biweekly random urine screenings, and monthly individual therapy sessions. The investigators will piggy-back off this existing structure and randomize Veterans with stimulant use disorders and receiving MMT for co-occurring OUD to receive either oxytocin or placebo, to be administered twice daily for six weeks while in the MMT program.
  Intranasal oxytocin: Each Veteran with a stimulant use disorder, receiving MMT for OUD will receive a oxytocin nasal spray 40IU to be self administered twice daily over 6 weeks while in the MMT program. The veteran will come in for a total of 7 weekly visits. At baseline and during the last visit the veteran will complete at Trier Social Stress Test (TSST), and psychophysiological and biomarkers of stress will be collected. At every weekly visit a urine sample and self-reported drug use will be collected and therapy attendance will be recorded.
Period: Overall Study
Arm/Group | Oxytocin | Placebo
Started | 18 | 22
Completed | 18 | 20
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Oxytocin: Oxytocin, to be administered intranasally twice daily for six weeks. TSST will be conducted prior to study drug administration and after the 6-week course.
- Placebo: Placebo, to be administered intranasally twice daily for six weeks. TSST will be conducted prior to study drug administration and after the 6-week course.
- Total: Total of all reporting groups
Arm/Group | Oxytocin | Placebo | Total
Number analyzed (Participants) | 18 | 22 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 14 | 32
  >=65 years | 0 | 8 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.94444 (11.35767) | 63.13636 (7.265676) | 59 (10.30061)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 18 | 22 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 16 | 23
  White | 8 | 4 | 12
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 22 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Stimulant Positive Drug Screen
Description: Aim 1: To evaluate the effectiveness of intranasal oxytocin on reducing stimulant use.
Time Frame: Baseline, Visits 1-7, up to 7 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 18 | 20
Participants
  Stimulant Positive: Baseline | 9 | 12
  Stimulant Positive: Week 1 | 9 | 10
  Stimulant Postive: Week 2 | 10 | 11
  Stimulant Positive: Week 3 | 8 | 11
  Stimulant Positive: Week 4 | 8 | 12
  Stimulant Positive: Week 5 | 9 | 12
  Stimulant Positive: Week 6 | 9 | 11
  Stimulant Positive: Week 7 | 9 | 11

2. Secondary Outcome: Working Alliance Inventory (WAI)
Description: Aim 2: To evaluate the effectiveness of intranasal oxytocin on improving psychosocial treatment engagement (social support) as measured by the Working Alliance Inventory, an inventory of therapeutic alliance. The Working Alliance Inventory is a 36 question inventory. Each item is scored from 1-7, minimum = 1 and maximum = 7. Minimum total score = 36 to maximum total score = 252. Higher scores represent higher satisfaction.
Time Frame: Visits 1 and 7, Up to 7 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 18 | 20
score on a scale
  WAI Week 1: Self-Report | 3.5972 (0.8816) | 3.8182 (0.8107)
  WAI Week 7: Self-Report | 3.4676 (0.785) | 3.5208 (1.0516)
  WAI Week 1:Therapist | 4.088 (0.7048) | 3.754 (0.7370)
  WAI Week 7: Therapist | 4.1450 (0.7334) | 3.7486 (0.8308)

3. Secondary Outcome: Heart Rate in Response to Trier Social Stress Test (TSST).
Description: Aim 3: To evaluate the effectiveness of intranasal oxytocin on reducing stress-related psycho-physiological measures in response to the Trier Social Stress Test (TSST).
  The Trier Social Stress Test is a series of tasks which predictably induce stress in participants. First, physiological states are measured at baseline. Then participants are told they must prepare a 5 minute speech for a panel of researchers, which they then present. Participants are then asked verbal arithmetic questions. Finally, this is followed by a period of 5 minute rest referred to as the 'cooldown' period.
  Heart rate was assessed at different time points during the TSST. These time point are as follows: baseline, during speech preparation, during speech presentation, during arithmetic problems, and during the cooldown period. Higher scores indicate higher stress levels.
Time Frame: Visits 1 and 7, up to 7 weeks
Measure: Mean (Standard Deviation); unit: Beats/minute
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 18 | 20
Beats/minute
  Heart Rate Baseline: Week 1 | 77.252 (8.34820) | 68.1912 (13.9445)
  Heart Rate During Speech Prep: Week 1 | 77.5306 (11.1108) | 69.8634 (13.2503)
  Heart Rate During Speech: Week 1 | 85.3146 (12.1203) | 79.4769 (15.1165)
  Heart Rate During Arithmetic: Week 1 | 85.1227 (10.65619) | 77.8194 (15.6546)
  Heart Rate Cooldown: Week 1 | 72.0023 (18.7152) | 68.8551 (12.1091)
  Heart Rate Baseline: Week 7 | 76.116 (8.7493) | 72.6821 (11.9550)
  Heart Rate During Speech Prep: Week 7 | 74.9320 (8.4512) | 69.9714 (12.1507)
  Heart Rate During Speech: Week 7 | 81.8189 (8.1597) | 79.2512 (14.2214)
  Heart Rate During Arithmetic: Week 7 | 82.6265 (8.4639) | 82.8517 (18.0291)
  Heart Rate Cooldown: Week 7 | 74.9591 (9.8852) | 68.8543 (11.8623)

4. Secondary Outcome: Respiratory Rate in Response to Trier Social Stress Test (TSST).
Description: Aim 3: To evaluate the effectiveness of intranasal oxytocin on reducing stress-related psycho-physiological measures in response to the Trier Social Stress Test (TSST).
  The Trier Social Stress Test is a series of tasks which predictably induce stress in participants. First, physiological states are measured at baseline. Then participants are told they must prepare a 5 minute speech for a panel of researchers, which they then present. Participants are then asked verbal arithmetic questions. Finally, this is followed by a period of 5 minute rest referred to as the 'cooldown' period.
  Respiratory rate was assessed at different time points during the TSST. These time point are as follows: baseline, during speech preparation, during speech presentation, during arithmetic problems, and during the cooldown period. Higher scores indicate higher stress levels.
Time Frame: Visits 1 and 7, up to 7 weeks
Measure: Mean (Standard Deviation); unit: Breaths/minute
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 18 | 20
Breaths/minute
  Respiratory Rate Baseline: Week 1 | 10.9117 (1.5119) | 11.2000 (2.9642)
  Respiratory Rate During Speech Prep: Week 1 | 11.0512 (3.3724) | 12.292 (2.9966)
  Respiratory Rate During Speech: Week 1 | 11.4533 (2.976) | 12.3352 (2.9521)
  Respiratory Rate During Arithmetic: Week 1 | 10.56 (1.7841) | 11.7565 (3.5337)
  Respiratory Rate Cooldown: Week 1 | 10.6278 (3.0036) | 10.5266 (2.1028)
  Respiratory Rate Baseline: Week 7 | 11.6779 (3.795) | 11.4583 (2.3595)
  Respiratory Rate During Speech Prep: Week 7 | 10.6251 (1.8414) | 12.7914 (3.7546)
  Respiratory Rate During Speech: Week 7 | 10.6675 (3.0857) | 11.5526 (3.304)
  Respiratory Rate During Arithmetic: Week 7 | 10.4215 (1.9839) | 12.4459 (2.4201)
  Respiratory Rate Cooldown: Week 7 | 9.9913 (2.6662) | 10.3816 (2.9001)

5. Secondary Outcome: Respiratory Sinus Arrythmia (RSA) in Response to Trier Social Stress Test (TSST).
Description: Aim 3: To evaluate the effectiveness of intranasal oxytocin on reducing stress-related psycho-physiological measures in response to the Trier Social Stress Test (TSST).
  The Trier Social Stress Test is a series of tasks which predictably induce stress in participants. First, physiological states are measured at baseline. Then participants are told they must prepare a 5 minute speech for a panel of researchers, which they then present. Participants are then asked verbal arithmetic questions. Finally, this is followed by a period of 5 minute rest referred to as the 'cooldown' period.
  Respiratory sinus arrythmia (RSA) was assessed at different time points during the TSST. These time point are as follows: baseline, during speech preparation, during speech presentation, during arithmetic problems, and during the cooldown period. Higher scores indicate higher stress levels.
Time Frame: Visits 1 and 7, up to 7 weeks
Measure: Mean (Standard Deviation); unit: milliseconds squared
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 18 | 20
milliseconds squared
  Respiratory Sinus Arrythmia During Baseline: Week 1 | 4.2435 (1.2701) | 4.9543 (1.8461)
  Respiratory Sinus Arrythmia During Speech Prep: Week 1 | 4.6264 (1.2903) | 4.7393 (1.5292)
  Respiratory Sinus Arrythmia During Speech: Week 1 | 3.5542 (1.2285) | 3.8212 (1.3293)
  Respiratory Sinus Arrythmia During Arithmetic: Week 1 | 3.5364 (1.1521) | 3.7893 (1.1818)
  Respiratory Sinus Arrythmia During Cooldown: Week1 | 4.3466 (1.0783) | 4.4933 (1.3137)
  Respiratory Sinus Arrythmia During Baseline: Week 7 | 4.1866 (1.1912) | 4.053 (1.7715)
  Respiratory Sinus Arrythmia During Speech Prep: Week 7 | 4.0099 (1.3911) | 4.2972 (1.6850)
  Respiratory Sinus Arrythmia During Speech: Week 7 | 3.6254 (1.3660) | 3.5998 (1.523)
  Respiratory Sinus Arrythmia During Arithmetic: Week 7 | 3.4825 (1.3147) | 3.5267 (1.3283)
  Respiratory Sinus Arrythmia During Cooldown: Week 7 | 3.9752 (1.4793) | 4.1651 (1.5196)

6. Secondary Outcome: Root Mean Square of Successive Differences (RMSSD) of Heart Rate Variability in Response to Trier Social Stress Test (TSST).
Description: Aim 3: To evaluate the effectiveness of intranasal oxytocin on reducing stress-related psycho-physiological measures in response to the Trier Social Stress Test (TSST).
  The Trier Social Stress Test is a series of tasks which predictably induce stress in participants. First, physiological states are measured at baseline. Then participants are told they must prepare a 5 minute speech for a panel of researchers, which they then present. Participants are then asked verbal arithmetic questions. Finally, this is followed by a period of 5 minute rest referred to as the 'cooldown' period.
  The root mean square of successive differences (RMSSD) were assessed at different time points during the TSST. These time point are as follows: baseline, during speech preparation, during speech presentation, during arithmetic problems, and during the cooldown period. Higher scores indicate higher stress levels. Calculated by measuring each successive time difference between heartbeats in ms.
Time Frame: Visits 1 and 7, up to 7 weeks
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 18 | 20
milliseconds
  RMSSD During Baseline: Week 1 | 26.8196 (41.5701) | 48.865 (48.2147)
  RMSSD During Speech Prep: Week 1 | 28.5447 (38.5287) | 37.7607 (44.6989)
  RMSSD During Speech: Week 1 | 22.5526 (44.3238) | 20.9388 (21.2336)
  RMSSD During Arithmetic: Week 1 | 21.113 (39.3470) | 21.1729 (18.4126)
  RMSSD During Cooldown: Week 1 | 29.7325 (53.4858) | 34.5220 (43.9497)
  RMSSD During Baseline Week 7 | 15.7941 (9.0513) | 26.3299 (30.7912)
  RMSSD During Speech Prep: Week 7 | 16.0198 (9.2258) | 28.1708 (31.7601)
  RMSSD During Speech: Week 7 | 12.9299 (7.5432) | 22.1121 (30.6961)
  RMSSD During Arithmetic: Week 7 | 11.3174 (6.5779) | 21.2057 (32.3207)
  RMSSD During Cooldown: Week 7 | 17.9728 (13.0228) | 24.6587 (20.8481)

7. Secondary Outcome: Self-reported Stimulant Craving
Description: Aim 4: To evaluate the effectiveness of intranasal oxytocin on reducing stimulant craving in response the Trier Social Stress Test (TSST).
  The Cocaine Craving Questionnaire (CCQ) (brief) was modified to include all stimulants and administered. The CCQ is a 10-item questionnaire, with each item ranking on a scale of 1-7. 1 indicates 'Strongly Disagree' and 7 indicates 'Strongly Agree'. Higher scores indicate higher rates of craving. The CCQ was administered at three distinct time points: before the TSST, immediately after the TSST and 20 minutes post-TSST.
  The Trier Social Stress Test is a series of tasks which predictably induce stress in participants. First, physiological states are measured at baseline. Then participants are told they must prepare a 5 minute speech for a panel of researchers, which they then present. Participants are then asked verbal arithmetic questions. Finally, this is followed by a period of 5 minute rest referred to as the 'cooldown' period.
Time Frame: Visits 1 and 7, Up to 7 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 18 | 20
score on a scale
  Pre_Trier: Week 1 | 2.1667 (1.1827) | 1.82727 (1.1707)
  Imm_Post_Trier: Week 1 | 2.4389 (1.7446) | 2.35 (1.6964)
  20m_Post_Trier: Week 1 | 2.3056 (1.4941) | 1.8955 (1.2688)
  Pre_Trier: Week 7 | 1.7167 (1.0755) | 1.42 (0.7135)
  Imm_Post_Trier: Week 7 | 1.6833 (0.8535) | 1.48 (0.818)
  20m_Post_Trier: Week 7 | 1.7167 (1.058) | 1.67 (1.0255)

8. Secondary Outcome: Individual and Group Therapy Attendance Rates
Description: Aim 5: To evaluate the effectiveness of intranasal oxytocin on improving psychosocial treatment engagement (social support) as measured by individual and group therapy attendance rates.
Time Frame: Visits 1-7, Up to 7 weeks
Measure: Mean (Standard Deviation); unit: proportion of OTP visits attended
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 18 | 20
proportion of OTP visits attended
  Attendance Proportion: Week 1 | 0.9352 (0.1416) | 0.8406 (0.3047)
  Attendance Proportion: Week 2 | 0.9333 (0.1183) | 0.8485 (0.2951)
  Attendance Proportion: Week 3 | 0.9241 (0.1652) | 0.8429 (0.3022)
  Attendance Proportion: Week 4 | 0.9260 (0.1828) | 0.7857 (0.3580)
  Attendance Proportion: Week 5 | 0.8704 (0.2181) | 0.7476 (0.3572)
  Attendance Proportion: Week 6 | 0.9444 (0.1560) | 0.7483 (0.3915)
  Attendance Proportion: Week 7 | 1 (0) | 0.75 (0.4443)

9. Secondary Outcome: Cortisol Levels in Response to Trier Social Stress Test (TSST).
Description: Aim 6: To evaluate the effectiveness of intranasal oxytocin on reducing stress biomarkers in response to the TSST.
Time Frame: Visits 1 and 7, up to 7 weeks
Measure: Mean (Standard Deviation); unit: (ug/dL)
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 18 | 20
(ug/dL)
  Initial Cortisol Levels (ug/dL) Week 1 | 0.331 (0.263) | 0.319 (0.335)
  Pre-Trier Cortisol Levels (ug/dL) Week 1 | 0.283 (0.213) | 0.193 (0.163)
  Immediately Post-Trier Cortisol Levels (ug/dL) Week 1 | 0.286 (0.221) | 0.242 (0.286)
  20Minutes Post-Trier Cortisol Levels (ug/dL) Week 1 | 0.29 (0.184) | 0.211 (0.245)
  Initial Cortisol Levels (ug/dL) Week 7 | 0.206 (0.155) | 0.259 (0.154)
  Pre-Trier Cortisol Levels (ug/dL) Week 7 | 0.156 (0.093) | 0.197 (0.115)
  Immediately Post-Trier Cortisol Levels (ug/dL) Week 7 | 0.167 (0.112) | 0.184 (0.09)
  20 Minutes Post-Trier Cortisol Levels (ug/dL) Week 7 | 0.175 (0.130) | 0.168 (0.073)

10. Secondary Outcome: Dehydroepiandrosterone (DHEA) Levels in Response to Trier Social Stress Test (TSST)
Description: Aim 6: To evaluate the effectiveness of intranasal oxytocin on reducing stress biomarkers in response to the TSST.
Time Frame: Visits 1 and 7, up to 7 weeks
Measure: Mean (Standard Deviation); unit: (pg/mL)
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 18 | 20
(pg/mL)
  Initial DHEA Levels (pg/mL) Week 1 | 86.230 (52.999) | 62.695 (67.462)
  Pre-Trier DHEA Levels (pg/mL) Week 1 | 90.313 (80.944) | 52.32 (55.91)
  Immediately Post-Trier DHEA Levels (pg/mL) Week 1 | 100.468 (76.830) | 63.471 (57.251)
  20 Minutes Post-Trier DHEA Levels (pg/mL) Week 1 | 81.742 (68.051) | 54.816 (52.980)
  Initial DHEA Levels(pg/mL) Week 7 | 87.674 (78.363) | 61.581 (77.382)
  Pre-Trier DHEA Levels (pg/mL) Week 7 | 75.221 (80.167) | 54.324 (57.183)
  Immediately Post-Trier DHEA Levels (pg/mL) Week 7 | 84.230 (72.875) | 69.291 (108.134)
  20 Minutes Post-Trier DHEA Levels (pg/mL) Week 7 | 82.009 (86.669) | 66.736 (103.362)

11. Secondary Outcome: Self-reported Stress/Anxiety
Description: Aim 7: To evaluate the effectiveness of intranasal oxytocin on reducing self-reported stress/anxiety levels in response to the TSST. The scale used to measure anxiety was the State-Trait Anxiety Inventory (STAI-6). This scale consists of 40 questions, all of which are rated on a 4-point likert scale. 1 indicates 'Almost Never' while 4 indicates 'Almost Always'. The minimum score is 0, indicating no anxiety, and maximum score is 63, indicating severe anxiety.
Time Frame: Visits 1 and 7, Up to 7 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 18 | 20
score on a scale
  Pre_Trier: Week 1 | 34.815 (13.778) | 32.2727 (11.0978)
  Imm_Post_Trier: Week 1 | 46.4815 (15.529) | 46.0606 (19.29)
  20m_Post_Trier: Week 1 | 36.8519 (14.4834) | 36.97 (14.5809)
  Pre_Trier: Week 7 | 35.185 (12.379) | 29.17 (11.38)
  Imm_Post_Trier: Week 7 | 42.222 (15.966) | 36.5 (11.7217)
  20m_Post_Trier: Week 7 | 35.741 (11.871) | 31 (11.726)

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Oxytocin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/22
Other Adverse Events (participants affected / at risk) | 1/18 | 1/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxytocin (N=18) | Placebo (N=22)
Constipation (Gastrointestinal disorders) | 1 (2) | 0 (0) — Participant (Subject Identifier (ID)# 730) was admitted to the San Francisco Veteran Affairs (SFVA) ER for constipation on 3/30/2019 and 4/10/2019. He was discharged on the same day for both events.
Stinging sensation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Participant (Subject ID# 730) reported a stinging sensation and was examined by study physician, who did not observe irritation. Participant said sensation subsided, and remarked. 'It must've been a zit'.
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1) — Participant (Subject ID# 731) reported dream-like hallucination that subsided after 2 seconds. Participant reported methamphetamine use prior to hallucination, and the event did not result in participant injury.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT03016598/Prot_000.pdf
  • Statistical Analysis Plan (2016-03-02): https://cdn.clinicaltrials.gov/large-docs/98/NCT03016598/SAP_001.pdf
  • Informed Consent Form (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/98/NCT03016598/ICF_002.pdf